CLINICAL TRIAL: NCT07293377
Title: Prospective Validation of a Risk Stratification Model for Mortality Up to 30 Days After Surgery
Brief Title: Prospective Validation of ExCARE Model for 30-Day Postoperative Mortality
Acronym: ExCARE-HNSC
Status: Completed | Type: Observational
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Andre Prato Schmidt, Associate Professor, Hospital Nossa Senhora da Conceicao
Other Study IDs: 56209622.5.0000.5530; Secondary ID 1: 5.507.979 (Other: Hospital Nossa Senhora da Conceicao)
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Complications
Keywords: Surgical Procedures; Mortality; Postoperative Care; Risk Assessment; Surgery; Anesthesia; Perioperative Medicine; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Patients Cohort: Adult patients (>18 years) undergoing elective, urgent, or emergency non-cardiac surgeries (excluding diagnostic procedures, sedation-only, local anesthesia, hepatic/pulmonary/cardiac transplants, or brain-dead organ donors). No intervention; routine care with prospective data collection.

SUMMARY:
This prospective observational cohort study aims to validate the ExCARE risk model, derived from four preoperative variables (age, ASA-PS classification, procedure urgency, and surgical magnitude), for predicting in-hospital mortality up to 30 days post-non-cardiac surgery in a Brazilian tertiary hospital. A secondary validation of the SORT (Surgical Outcome Risk Tool) model will also be performed for comparison. The study involves no interventions and focuses on risk stratification to improve perioperative care allocation.

DETAILED DESCRIPTION:
Approximately 300 million major surgical procedures are performed worldwide annually, with postoperative complications increasing costs and mortality. This study addresses the need for better perioperative risk stratification in Brazil, following WHO recommendations for universal health coverage. The ExCARE model, developed from 13,581 patients at Hospital de Clínicas de Porto Alegre (HCPA), showed good discriminative capacity (repeated in a 7,254-patient validation cohort). This external prospective validation at Hospital Nossa Senhora da Conceição will assess its performance in a new setting. Patients are stratified into four risk classes: Class I (<2% mortality), Class II (2-5%), Class III (5-10%), Class IV (>10%). Data will be analyzed using logistic regression, AUROC for discrimination, and Hosmer-Lemeshow test for calibration. Expected enrollment: 3,000 patients over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years; Scheduled for elective, urgent, or emergency surgeries at Hospital Nossa Senhora da Conceição; For multiple surgeries in one admission, only the major procedure considered.

Exclusion Criteria:

* Diagnostic procedures; Sedation-only or local anesthesia; Hepatic, pulmonary, or cardiac transplants; Brain-dead patients for organ donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this prospective observational cohort study consists of adult patients aged over 18 years who are scheduled for elective, urgent, or emergency non-cardiac surgeries at the Hospital Nossa Senhora da Conceição in Porto Alegre, Brazil. Patients are recruited via convenience sampling from those routinely attending the hospital's surgical center and meeting the inclusion criteria.
  Key inclusion criteria:
  Age greater than 18 years. Undergoing elective, urgent, or emergency surgical procedures.
  Key exclusion criteria:
  Patients scheduled for diagnostic procedures. Procedures performed under sedation only or local anesthesia. Patients undergoing hepatic, pulmonary, or cardiac transplants. Patients diagnosed with brain death and undergoing organ donation. In cases of multiple surgical interventions during the same hospitalization, only the procedure of greatest magnitude is considered for outcome analysis.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality within 30 days post-surgery | 30 days
  In-hospital mortality within 30 days post-surgery (Time Frame: 30 days; Measured as binary outcome: death [1] or discharge/alive [0]; Analyzed via ExCARE model probability and logistic regression)

SECONDARY OUTCOMES:
Performance of SORT model for 30-day mortality prediction | 30 days
  Performance of SORT model for 30-day mortality prediction (Time Frame: 30 days; Compared to ExCARE via AUROC, calibration, and risk ratios)

CONTACTS AND LOCATIONS:
Overall Officials: Andre P. Schmidt, MD, PhD, Principal Investigator — Hospital Nossa Senhora da Conceição
Locations (1):
- Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Size and distribution of the global volume of surgery in 2012. Bull World Health Organ. 2016 Mar 1;94(3):201-209F. doi: 10.2471/BLT.15.159293. PMID 26966331
- [Result] Moonesinghe SR, Mythen MG, Das P, Rowan KM, Grocott MP. Risk stratification tools for predicting morbidity and mortality in adult patients undergoing major surgery: qualitative systematic review. Anesthesiology. 2013 Oct;119(4):959-81. doi: 10.1097/ALN.0b013e3182a4e94d. PMID 24195875
- [Result] Protopapa KL, Simpson JC, Smith NC, Moonesinghe SR. Development and validation of the Surgical Outcome Risk Tool (SORT). Br J Surg. 2014 Dec;101(13):1774-83. doi: 10.1002/bjs.9638. PMID 25388883
- [Result] Gutierrez CS, Passos SC, Castro SMJ, Okabayashi LSM, Berto ML, Lorenzen MB, Caumo W, Stefani LC. Few and feasible preoperative variables can identify high-risk surgical patients: derivation and validation of the Ex-Care risk model. Br J Anaesth. 2021 Feb;126(2):525-532. doi: 10.1016/j.bja.2020.09.036. Epub 2020 Oct 27. PMID 33127046
- [Result] Stefani LC, Gutierrez CS, Castro SMJ, Zimmer RL, Diehl FP, Meyer LE, Caumo W. Derivation and validation of a preoperative risk model for postoperative mortality (SAMPE model): An approach to care stratification. PLoS One. 2017 Oct 30;12(10):e0187122. doi: 10.1371/journal.pone.0187122. eCollection 2017. PMID 29084236